CLINICAL TRIAL: NCT00326404
Title: Continuous Versus Cyclic Use of an Oral Contraceptive Pills in Adolescents
Brief Title: Continuous Versus Cyclic Use of Oral Contraceptive Pills in Adolescents
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Lisa Allen/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000008437
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Contraception
Keywords: Oral Contraceptives; Adolescents; Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Desogestrel-Ethinyl Estradiol 21 tablets
- 2 (Active Comparator)
  Interventions: Drug: Desogestrel-Ethinyl Estradiol 28 tablets

INTERVENTIONS:
Drug: Desogestrel-Ethinyl Estradiol 21 tablets — The participants in the continuous study arm will be given 4 packs of Marvelon-21, so that they can take the pills continuously for 84 days followed by no medication for 7 days. During these 7 days, the participant will have a withdrawal bleed. This sequence is repeated by the participant for a total of 12 months. Each patient in the continuous arm will have 4 withdrawal bleeds per year.
  Other Names: Marvelon-21
  Arms: 1
Drug: Desogestrel-Ethinyl Estradiol 28 tablets — The participants in the cyclical arm of the study will be given 3 packs of Marvelon-28 and asked to take all the pills in the packet, including the placebo pills. During the week of placebo pills, these participants will have a withdrawal bleed. Each patient in the cyclical arm will have 12 withdrawal bleeds per year. The duration of study drug treatment for both arms is 12 months.
  Other Names: Marvelon-28
  Arms: 2

SUMMARY:
The primary purpose of this study is to compare the compliance rates of adolescents who take oral contraceptives (OCPs) continuously to those who take OCPs cyclically.

DETAILED DESCRIPTION:
Oral contraceptive pills have traditionally been prescribed in a cyclical manner, where there are 21-24 days of active pills and 4-7 days of placebo pills or a pill-free interval, creating a 28-day cycle. It has now been proven that as long as a woman has both estrogen and progesterone, her uterine lining is protected and is thin. To that effect, a new OCP (Seasonale®, Barr Laboratories, Pomona, NY) has been packaged in the United States that combines 84 days of active pills with 7 days of placebo pills. This allows a withdrawal bleed every 3 months.

Like in adult women, OCPs are the most popular form of birth control and cycle control in adolescents. But, for a variety of reasons, adolescents tend to have poorer compliance when taking OCPs. Adult women tend to be noncompliant about 6% of the time, but, by the end of one year, adolescents have a non-compliance rate of 34-66%.

There have been few studies that even describe improved compliance and decreased ovarian follicular development in women who take OCPs continuously, which could be beneficial in decreasing the rate of adolescent pregnancy. The majority of the studies looking at continuous use of OCPs have been performed in adult women. At present, there has been only one article that has addressed the use of continuous OCPs in adolescents. Sucato and Gold discussed the indications of continuous use of OCPs, how to prescribe them, and what type of progestin to use; but they did not specifically examine compliance or the safety and efficacy of continuous OCPs in adolescents. We plan to evaluate these issues in our study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 15 to 18
* Presenting to the Gynecology and Adolescent Medicine Clinic for contraception

Exclusion Criteria:

* Prior use of the study medication with no improvement in symptoms
* Any medical condition that indicates continuous OCPs (i.e. acute menorrhagia, dysmenorrhea that did not previously respond to cyclical OCP use)
* Personal history of or current thromboembolic disorder
* First-degree relative(s) with thromboembolic disorder
* Cerebrovascular disease
* Coronary artery disease
* Cardiac valvular disease
* Hypertension (systolic blood pressure > 160 mmHg or diastolic > 100 mmHG)
* Diabetes with retinopathy/neuromyopathy/nephropathy)
* Breast cancer
* Endometrial cancer
* Undiagnosed abnormal uterine bleeding
* Cholestatic jaundice of pregnancy
* Hepatic tumor
* Known or suspected pregnancy
* Less than 6 months postpartum if breastfeeding
* Classic migraine with aura or any other neurological signs
* Gallbladder disease
* Taking any medications known to affect the efficacy of OCPs (i.e. phenytoin, phenobarbital, primidone, carbamazepine, griseofulvin, rifampin)

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare the compliance rates of adolescents who take OCPs continuously to those who take OCPs cyclically. | 1 year

SECONDARY OUTCOMES:
The number of girls who have positive pregnancy test results at 12 months | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Allen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Walpole B, Dettmer E, Morrongiello B, McCrindle B, Hamilton J. Motivational interviewing as an intervention to increase adolescent self-efficacy and promote weight loss: methodology and design. BMC Public Health. 2011 Jun 10;11:459. doi: 10.1186/1471-2458-11-459. PMID 21663597